CLINICAL TRIAL: NCT00607035
Title: The Japan-Combined Treatment With Olmesartan and a Calcium Channel Blocker Versus Olmesartan and Diuretics Randomized Efficacy Study (J-CORE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jichi Medical University (Other)
Responsible Party: Kazuomi Kario, Jichi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J_Core_071226; J_Core_071226_01
Record Dates: First submitted 2007-12-26; First posted 2008-02-05 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): The ARB plus CCB combination therapy group is administered olmesartan 20 mg/day and azelnidipine 16 mg/day for 6 months.
  Interventions: Drug: Olmesartan medoxomil ＋Azelnidipine
- H (Experimental): The ARB plus Diuretics combination therapy group is administered olmesartan medoxomil 20mg/day and hydrochlorothiazide 12.5mg/day for 6 months.
  Interventions: Drug: Olmesartan medoxomil + Hydrochlorothiazide

INTERVENTIONS:
Drug: Olmesartan medoxomil ＋Azelnidipine — The ARB plus CCB combination therapy group is administered olmesartan 20 mg/day and azelnidipine 16 mg/day for 6 months.
  Other Names: arm A
  Arms: A
Drug: Olmesartan medoxomil + Hydrochlorothiazide — The ARB plus Diuretics combination therapy group is administered olmesartan medoxomil 20mg/day and hydrochlorothiazide 12.5mg/day for 6 months.
  Other Names: arm H
  Arms: H

SUMMARY:
The purpose of this study is to investigate which combination therapy is more effective for improving the blood pressure (BP) and reducing target organ damage in Japanese hypertensive patients: Angiotensin II receptor blocker (ARB) plus calcium channel blocker (CCB) or ARB plus diuretics.

DETAILED DESCRIPTION:
Renin-angiotensin (RA) inhibitors have been demonstrated to be the most effective drugs for reducing subclinical target organ damage in hypertensive patients. In several patients, however, BP control is not sufficiently achieved by RA inhibitors alone, and a combination of two drugs is frequently required. It is unclear whether a combination of RA inhibitors and diuretics or CCB is more effective in reducing hypertensive target organ damage. Control of central BP has been shown to be more effective than peripheral BP in predicting cardiovascular events and target organ damage associated with hypertension. The J-CORE study is active controlled, 2-arm parallel group comparison, prospective randomized open blinded end-point (PROBE) design study. The ARB plus CCB combination therapy group is administered olmesartan 20 mg/day and azelnidipine 16 mg/day and the ARB plus diuretics combination therapy group receives olmesartan 20 mg/day and hydrochlorothiazide (HCTZ) 12.5 mg/day. At least 100 patients will be enrolled in each group and the follow up duration will be 24 weeks. The primary endpoint is to compare the changes in the central aortic BP and the ambulatory BP between the two groups. The secondary endpoint is to compare the changes in office BP, home BP, and hypertensive target organ damage between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive outpatients aged 30 years or older, and less than 85 years (at the time of informed consent), regardless of sex
* Office systolic BP/diastolic BP > 140/90 mmHg in a sitting position even if on treatment with olmesartan 20 mg/day for 3 months.

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* History of myocardial infarction or cerebrovascular accidents within 6 months prior to the screening
* Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass grafting (CABG) done within 6 months of screening or scheduled
* Current treatment for congestive cardiac failure (New York Heart Association [NYHA] functional class II or severer) or ejection fraction <40%
* Atrial fibrillation or atrial flutter
* Renal dysfunction (serum creatinine ≥2 mg/dl)
* Hepatic dysfunction (AST and/or ALT ≥100 IU/l)

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Changes in central BP and ambulatory BP | 6 months

SECONDARY OUTCOMES:
Changes in office BP and home BP. | 6 months
Changes in hypertensive target organ damage. Clinical laboratory data. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, Principal Investigator — Jichi Medical University School of Medicine
Locations (1):
- Jichi Medical University School of Medicine, Tochigi, Japan

REFERENCES:
- [Derived] Matsui Y, O'Rourke MF, Hoshide S, Ishikawa J, Shimada K, Kario K. Combined effect of angiotensin II receptor blocker and either a calcium channel blocker or diuretic on day-by-day variability of home blood pressure: the Japan Combined Treatment With Olmesartan and a Calcium-Channel Blocker Versus Olmesartan and Diuretics Randomized Efficacy Study. Hypertension. 2012 Jun;59(6):1132-8. doi: 10.1161/HYPERTENSIONAHA.111.189217. Epub 2012 Apr 30. PMID 22547439
- [Derived] Matsui Y, Eguchi K, O'Rourke MF, Ishikawa J, Shimada K, Kario K. Association between aldosterone induced by antihypertensive medication and arterial stiffness reduction: the J-CORE study. Atherosclerosis. 2011 Mar;215(1):184-8. doi: 10.1016/j.atherosclerosis.2010.12.022. Epub 2010 Dec 30. PMID 21241987
- [Derived] Matsui Y, Eguchi K, O'Rourke MF, Ishikawa J, Miyashita H, Shimada K, Kario K. Differential effects between a calcium channel blocker and a diuretic when used in combination with angiotensin II receptor blocker on central aortic pressure in hypertensive patients. Hypertension. 2009 Oct;54(4):716-23. doi: 10.1161/HYPERTENSIONAHA.109.131466. Epub 2009 Aug 10. PMID 19667251